CLINICAL TRIAL: NCT03332043
Title: High-resolution, Relational, Resonance-based, Electroencephalic Mirroring (HIRREM) for Pre-Hypertension: A Randomized, Controlled Clinical Trial
Brief Title: HIRREM for Pre-Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pre-hypertension no longer exists
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00044598
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Prehypertension; Blood Pressure; Autonomic Nervous System Imbalance; Cardiovascular Risk Factor; Cardiovascular Diseases; Brain Diseases
Keywords: HIRREM; Neurotechnology; Closed-loop; Acoustic stimulation; Allostatic; Heart rate variability; Baroreflex sensitivity; Blood pressure management; Autocalibration; Neural oscillations; Relaxation; Electroencephalic
MeSH Terms: conditions — Prehypertension; Cardiovascular Diseases; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- HIRREM (Experimental): Subjects in the experimental arm will receive an in-office, open-label course of acoustic stimulation linked to brain activity (High-resolution, relational, resonance-based, electroencephalic mirroring, HIRREM).
  Interventions: Device: HIRREM
- Ambient Nature Sounds (Active Comparator): Subjects in the active comparator arm will receive an in-office, open-label course of acoustic stimulation not linked to brain activity (ambient natures sounds).
  Interventions: Other: Ambient Nature Sounds

INTERVENTIONS:
Device: HIRREM — HIRREM (Brain State Technologies, Scottsdale, AZ) is a closed-loop, allostatic, acoustic stimulation neurotechnology that uses software-guided algorithmic analysis to identify and translate selected brain frequencies into audible tones of varying pitch and timing, to support real-time self-optimization of brain activity.
  Other Names: High-resolution, relational, resonance-based, electroencephalic mirroring
  Arms: HIRREM
Other: Ambient Nature Sounds — Digitally recordings of various ambient nature sounds such as a stream, waterfall, ocean waves, or rainfall, are provided via ear buds.
  Other Names: Wave Aid
  Arms: Ambient Nature Sounds

SUMMARY:
This randomized, controlled clinical pilot trial will evaluate the effects associated with in-office use of closed-loop, acoustic stimulation neurotechnology (High-resolution, relational, resonance-based, electroencephalic mirroring; HIRREM), compared with acoustic stimulation not linked to brainwaves (ambient nature sounds), for participants with pre-hypertension. Data collection will occur at baseline, and at intervals after completion of the intervention. Outcomes include blood pressure, measures of autonomic cardiovascular regulation, behavioral symptom outcomes, quality of life, alcohol use, and functional performance measures. The primary outcome will be change in blood pressure from baseline to 4-6 weeks after intervention.

DETAILED DESCRIPTION:
This will be a randomized, single site, controlled, pilot clinical trial, to evaluate the effects of in-office use of a closed-loop, allostatic, acoustic stimulation neurotechnology (High-resolution, relational, resonance-based, electroencephalic mirroring; HIRREM), compared with acoustic stimulation not linked to brainwaves (ambient nature sounds). Assuming a potential drop-out rate of 20%, up to 24 subjects will be enrolled to achieve a goal of having at least 20 subjects (10 per group) complete the study, per protocol. Patients who have blood pressures between 120-139 mm/Hg systolic, and/or 80-89 mm/Hg diastolic, as documented by their health care providers on two separate occasions, and no other exclusions, will be randomly assigned to receive either 8-16 sessions of either acoustic stimulation linked to brainwave activity (HCC), or acoustic stimulation not linked to brainwave activity (NCC), over a maximum of 4 weeks, with both groups continuing their current care throughout. There will be pre- and post-intervention data collection to include systolic and diastolic BP, and many secondary outcome measures including measures of autonomic cardiovascular regulation (continuous recording of BP and HR for calculation of measure of HRV and BRS), behavioral symptom outcomes (ISI, PSQI, ESS, CES-D, GAD-7, PCL-C, PSS), quality of life measure (QOLS), alcohol use (Audit C), and function performance measures (drop stick reaction testing, and grip strength). All measures will be collected at an enrollment visit (V1), and the intervention will begin 1-14 days later. BP and HR recordings will also be repeated prior to the start of the 7th session. Post-intervention data collections will be obtained at 1-7 days (V2), 4-6 weeks (V3, primary outcome), and 12-14 weeks (V4) following completion of the intervention. The primary outcome will be differential change in the systolic and diastolic BP from V1 to V3. Additional follow up (V4) will evaluate durability of effects. Following V4, those in the NCC group will be offered the opportunity to cross over to receive a course of HCC, and will continue to be followed for data collections at 1-7 days (V5), 4-6 weeks (V6), and 12-14 weeks (V7) after completing their crossover HCC sessions. Linear mixed models (LMMs) will be used to contrast longitudinal changes in systolic and diastolic blood pressure between the HCC and NCC groups. Mean contrasts will be used to compare the changes in blood pressures between groups from V1 to V3, our primary test of efficacy. Additional mean contrasts will be constructed to evaluate the consistency of any benefit of HIRREM through subsequent visits beyond V3. Comparisons of changes in all secondary outcomes will be assessed in a similar fashion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ≥ 18 years of age, with pre-hypertension, who have systolic BP ranging from 120-139 mm/Hg, or who have diastolic BP ranging from 80-89 mm/Hg.

Exclusion Criteria:

* Blood pressure values that are outside of the range for prehypertension at the enrollment visit.
* Unable, unwilling, or incompetent to provide informed consent.
* Physically unable to come to the study visits, or to sit comfortably in a chair for up to two hours at a time.
* Prior diagnosis of hypertension.
* Ongoing need for medical treatment for hypertension, or for the use of medications commonly used for treatment of hypertension.
* Known cardiovascular disease.
* Known seizure disorder.
* Known or anticipated pregnancy (females of childbearing age will be tested for pregnancy prior to randomization).
* Severe hearing impairment (because the subject will be using headphones during the interventions).
* Ongoing need for treatment with opiate, benzodiazepine, or anti-psychotic medications, anti-depressant medications such as SSRI, SNRI, or tricyclic, and sleep medications such as zolpidem or eszopiclone.
* Anticipated and ongoing use of recreational drugs, alcohol, or energy drinks
* Ongoing need for treatment with thyroid medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Data used for analysis of primary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  Change in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The severity of insomnia symptoms is measured using the ISI with each data collection visit. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28.
Pittsburgh Sleep Quality Index (PSQI) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The PSQI is a 19 item inventory that assesses sleep quality over a 1-month time interval. Items are weighted on a 0-3 interval scale. A global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Epworth Sleepiness Score (ESS) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The ESS measures a person's general level of daytime sleepiness, or their average sleep propensity in daily life. The simple questionnaire is based on retrospective reports of the likelihood of dozing off or falling asleep in a variety of different situations. Rated on a 4-point scale (0-3), it evaluates their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24.
Center for Epidemiologic Studies Depression Scale (CES-D) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a depression scale which will help to assess this co-morbidity. CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off.
Generalized Anxiety Disorder-7 (GAD-7) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The Generalized Anxiety Disorder-7 (GAD-7) is a seven item screening tool for anxiety that is widely used in primary care. GAD-7 is a brief, reliable and valid measure of assessing generalized anxiety disorder.
PTSD Checklist for Civilians (PCL-C) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The PTSD Checklist for civilians (PCL-C), measures the American Psychiatric Association's Diagnostic and statistical manual of mental disorders (DSM-IV) Criteria B, C, & D of PTSD symptoms based on traumatic life experience related to military service. Seventeen items are rated on a Likert scale with a composite score range of 17 to 85. A score of 44 or higher correlates with probability of civilian-related PTSD.
Perceived Stress Scale (PSS) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The Perceived Stress Scale (PSS) is a ten-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale, with answers rated from 0-4, also includes a number of direct queries about current levels of experienced stress.
Quality of Life Scale (QOLS) | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The Quality of Life Scale (QOLS) is a 16-item scale that was modified from a 15-item scale used in chronic disease patients. Topics include different components of daily life such as relationships, community engagement, personal fulfillment, and recreation. Each item is scaled from 1 to 7 and a sum score is calculated to represent higher levels of satisfaction in life (range is 16-112).
AUDIT-C | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  The AUDIT-C is a short, 3-item alcohol screening for hazardous drinkers or active alcohol use disorders. This measure consists of 3 questions to assess an individual's alcohol use. Each question has five possible answers ranging from of 0-4 with a total scoring scale of 0-12. A total score of 3 or more in women and a score of four or more in men is suggestive of hazardous drinking or active alcohol use disorders. This form is modified from the longer, 10-item AUDIT instrument.
Reaction Testing | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  Reaction testing will be evaluated by a drop-stick, clinical reaction time apparatus. It is constructed from a meter stick covered in friction tape with gradations. The modified meter stick is fixed to a weighted rubber cylinder. The apparatus is placed between the thumb and index finger of the subject and released at a random time during a countdown. The subject catches the apparatus and the distance fallen (cm) is converted to reaction. Following two practice trials, subjects perform eight trials, and a mean distance value is used for analysis. This is repeated with a second set of 8 trials later during the enrollment visit, and the mean distance value from the second trial will be used as the baseline value. Use of the average distance from the second set of trials will be used as the baseline value so as to avoid the impact of learning effect for this test.
Grip Strength | Data used for analysis of secondary outcome is collected at the enrollment visit, 1-7 days after the intervention is completed, 4-6 weeks after the intervention is completed, and 12-14 weeks after completion of the intervention
  Grip strength will be evaluated using a hydraulic hand dynamometer (Baseline Hydraulic Hand Dynamometer). The greatest force generated during three trials will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No
Data will be shared in publications and presentations. No plan to formally make individual participant data available for this study.

REFERENCES:
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- See also: HIRREM research webpage — http://wakehealth.edu/hirrem

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03332043/Prot_SAP_000.pdf